CLINICAL TRIAL: NCT01997749
Title: The Effect of a Ketogenic Diet on Blood Glucose, Function and Disease Progress in Acute Stroke Patients
Brief Title: Effects of a Ketogenic Diet on Acute Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Arne Astrup, Dr.Med.Sci./Ph.D., University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G-1-2013-012
Record Dates: First submitted 2013-10-28; First posted 2013-11-28 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Acute Stroke
Keywords: stroke, ketogenic diet, ketosis, ischemia, brain, ketones, hyperglycemia, neuroprotection
MeSH Terms: conditions — Stroke; Ketosis; Ischemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketogenic diet (Experimental): Acute stroke patients will receive a ketogenic diet (Ketocal 4:1 and ketogenic meals) for the first week after inclusion
  Interventions: Dietary Supplement: Ketocal 4:1 (Nutricia); Dietary Supplement: Ketogenic meals
- Control diet (Active Comparator): Acute stroke patients will receive a control diet (the regular diet, enteral or oral, offered at the hospitals) for the first week after inclusion.
  Interventions: Dietary Supplement: Control diet: Regular diet offered at the hospitals

INTERVENTIONS:
Dietary Supplement: Ketocal 4:1 (Nutricia)
  Arms: Ketogenic diet
Dietary Supplement: Control diet: Regular diet offered at the hospitals
  Arms: Control diet
Dietary Supplement: Ketogenic meals
  Arms: Ketogenic diet

SUMMARY:
The purpose of this controlled, randomized intervention is to investigate whether a fat-based (ketogenic) diet given for a week has a positive effect on blood sugar, mortality and function in patients hospitalized with acute stroke compared to the effect of a usual diet.

The study hypothesis is that a ketogenic diet and reduced availability of glucose to the brain cells will reduce the volume of neuronal damage in the brain and improve function.

The intervention will take place at the neurological units of Glostrup and Bispebjerg Hospital in Denmark.

DETAILED DESCRIPTION:
A ketogenic diet can induce ketosis after a period of 2-3 days and offer the brain an alternative energy substrate to glucose in the form of ketone bodies. Feeding the brain ketone bodies can potentially benefit a stroke patient's brain in several ways:

Stroke is characterized by impaired blood and oxygen supply to brain cells. This can cause glucose to convert to lactate which is toxic for the brain. Decreasing glucose availability to brain cells may thus potentially decrease the area of damage in the ischemic penumbra (perifephery of the stroke). Compared with sugar, burning ketone bodies requires less oxygen to produce the same amount of energy, suggesting that brain cells could have a potential greater chance of surviving during circumstances of reduced oxygen supply. By decreasing mitochondria activity, ROS synthesis is also decreased, which can help decrease the necrotic area around the ischemic penumbra. Furthermore, the ketogenic diet does not induce an increase in blood sugar which could be an advantage since many stroke patients are admitted with hyperglycemia associated with a worse outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic or hemorrhagic stroke.
* NIHSS score of at least 5.
* Both primary and recurrent cases.
* Inclusion as early as possible, but no later than 72 hours from symptom onset.
* Patients with expected hospitalization for a minimum of seven days.
* Adult patients with cognitive ability to give informed consent.
* Patients with writing and orally accepted participation.

Exclusion Criteria:

* Patients with SAH and traumatic hematoma.
* Patients with pancreatic insufficiency (steatorrhea).
* Patients unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline NIHSS (national institute of health stroke scale) at 90 days | Baseline and 90 days
  NIHSS is a common stroke scale used to objectively quantify the impairment caused by a stroke
Change from baseline fasting blood sugar at 7 days | Baseline and 7 days
Change from baseline p-C-peptide at 7 days | Baseline and 7 days

SECONDARY OUTCOMES:
Change from baseline p-triglyceride (fasting) at 7 days | Baseline and 7 days
Change from baseline p-LDL at 7 days | Baseline and 7 days
Change from baseline p-CRP at 7 days | Baseline and 7 days
Change from baseline p-beta-hydroxy butyrate at 7 days | Baseline and 7 days
Change from baseline p-phosphate at 7 days | Baseline and 7 days
Change from baseline p-potassium at 7 days | Baseline and 7 days
Change from baseline p-ALAT at 7 days | Baseline and 7 days
Change from baseline p-alkaline phosphatase at 7 days | baseline and 7 days
Change from baseline p-bilirubine at 7 days | baseline and 7 days
Change from baseline INR at 7 days | baseline and 7 days
Number of patients who died (mortality) | up to 3 months
Number of patients with pneunomia | Up to one week
Number of patients with gastrointestinal complications | Up to one week
  Gastrointestinal complications monitored daily are: Nausea, Vomiting, Constipation, Diarrhea, Abdominal pain
Change from baseline urine-ketones at 7 days | Baseline and 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Copenhagen, Denmark